CLINICAL TRIAL: NCT02793622
Title: Prevention of Malaria in HIV-uninfected Pregnant Women and Infants
Acronym: PROMOTE-BC3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Grant Dorsey, M.D, Ph.D., Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROMOTE-BC3
Record Dates: First submitted 2016-05-20; First posted 2016-06-08 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Malaria
Keywords: Chemoprevention; Malaria; Sulfadoxine-Pyrimethamine; Dihydroartemisinin-Piperaquine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy (Active Comparator): Women will be given SP (3 full strength tabs, 500 mg/25 mg) every four weeks times during pregnancy. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two drugs on day 1 (SP and placebo or DP and placebo) followed by one drug on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Interventions: Drug: Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy
- Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy (Active Comparator): Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) every 4 weeks during pregnancy. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two drugs on day 1 (SP and placebo or DP and placebo) followed by one drug on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Interventions: Drug: Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy

INTERVENTIONS:
Drug: Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy
  Other Names: Kamsidar (KPI)
  Arms: Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy
Drug: Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
  Other Names: Duo-Cotexin (Holley-Cotec)
  Arms: Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy

SUMMARY:
This will be a double-blinded randomized controlled phase III trial of 782 HIV uninfected pregnant women and the children born to them. HIV uninfected women at 12-20 weeks gestation will be randomized in equal proportions to one of two intermittent preventive treatment in pregnancy (IPTp) treatment arms: 1) monthly sulfadoxine-pyrimethamine (SP), or 2) monthly dihydroartemisinin-piperaquine (DP). Both interventions arms will have either SP or DP placebo to ensure adequate blinding is achieved in the study. Follow-up for the pregnant women will end approximately 6 weeks after giving birth. All children born to mothers enrolled in the study will be followed from birth until they reach 12 months of age.

DETAILED DESCRIPTION:
Pregnant women will be scheduled to be seen in the clinic every 4 weeks during their pregnancy and then 1 and 6 weeks following delivery. In addition, pregnant women will be instructed to come to the study clinic for all their medical care and avoid the use of any outside medications. Children will be scheduled to be seen in the clinic at 1, 4, 6, and 8 weeks of age and then every 4 weeks until they reach 52 weeks of age. Parents/guardians will be instructed to bring their children to the study clinic for all medical care and avoid the use of any outside medications. The study clinic will remain open 7 days a week from 8 a.m. to 5 p.m. Study participants not seen in the clinic for their every 4 week routine visits will be visited at home and requested to come to the study clinic as soon as possible. Pregnant women and children will receive standard of care as designated in the Uganda Ministry of Health guidelines. Routine antenatal care will include screening and treatment for sexually transmitted infections, blood pressure assessment, urine dipstick for proteinuria, prescription of iron, folate, multivitamins and mebendazole. Routine care in children will include immunizations, vitamin A supplementation, and management of anemia using Integrated Management of Childhood Illness (IMCI) guidelines. During routine assessments subjects will be asked about visits to outside health facilities and the use of any medications outside the study protocol. Standardized assessment of adherence will be done for study drugs administered at home and insecticide treated net use. A routine history and physical exam will be performed using a standardized clinical assessment form. Blood will be collected by finger prick for thick smear (in very young children, heel sticks may be substituted for finger pricks), capillary plasma (for routine visits where phlebotomy is not done in pregnant women only) and filter paper samples. If a pregnant woman or parent/guardian of a child reports a fever in the last 24 hours or the patient has a documented temperature > 38.0˚C tympanic, the patient's thick blood smear will be read immediately and if positive the patient will be diagnosed and treated for malaria. If the thick blood smear is negative, the patient will be managed by study physicians for a non-malarial febrile illness. If the patient is afebrile and does not report a recent fever, a thick blood smear will not be obtained, except when following routine testing schedules. In pregnant mothers, thick blood smears other than those done when a mother has fever will not be used for clinical care of study participants. Phlebotomy for routine laboratory tests (CBC and ALT) to monitor for potential adverse events from study medications, storage of plasma and for immunology studies will be performed every 8 weeks in pregnant women. Phlebotomy for routine laboratory tests (CBC) and immunology studies will be performed at 12, 28, and 52 weeks of age in children. For pregnant women, study drugs will be administered at the time of each routine visit. ECGs will be performed to measure the QTc interval in all pregnant women just prior to the 1st dose of study drugs and 2-3 hours after their 3rd dose of study drugs at 20, 28 and 36 weeks of gestation. In addition a finger prick capillary plasma sample will be collected just prior to performing the ECGs after the 3rd dose of study drugs at 20, 28, and 36 weeks of gestation in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy confirmed by positive urine pregnancy test or intrauterine pregnancy by ultrasound
* Estimated gestational age between 12-20 weeks
* Confirmed to be HIV uninfected by rapid test
* 16 years of age or older
* Resident of Busia District, Uganda
* Provision of informed consent by the pregnant woman for herself and her unborn child
* Agreement to come to the study clinic for any febrile episode or other illness and avoid medications given outside the study protocol
* Plan to deliver in the hospital

Exclusion Criteria:

* History of serious adverse event to SP or DP
* Active medical problem requiring inpatient evaluation at the time of screening
* Intention of moving outside of Busia District, Uganda
* Chronic medical condition requiring frequent medical attention
* Prior SP preventive therapy or any other antimalarial therapy during this pregnancy
* Early or active labor (documented by cervical change with uterine contractions)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Dorsey, MD PhD, Principal Investigator — University of California, San Francisco; Diane V Havlir, MD, Principal Investigator — University of California, San Francisco; Moses Kamya, MBChB MMed PhD, Principal Investigator — Makarere Univeritys ; Infectious Disease Research Collaboration
Locations (1):
- IDRC - Tororo Research Clinic, Tororo, Uganda

REFERENCES:
- [Result] Kajubi R, Ochieng T, Kakuru A, Jagannathan P, Nakalembe M, Ruel T, Opira B, Ochokoru H, Ategeka J, Nayebare P, Clark TD, Havlir DV, Kamya MR, Dorsey G. Monthly sulfadoxine-pyrimethamine versus dihydroartemisinin-piperaquine for intermittent preventive treatment of malaria in pregnancy: a double-blind, randomised, controlled, superiority trial. Lancet. 2019 Apr 6;393(10179):1428-1439. doi: 10.1016/S0140-6736(18)32224-4. Epub 2019 Mar 22. PMID 30910321
- [Result] Harrington WE, Kakuru A, Jagannathan P. Malaria in pregnancy shapes the development of foetal and infant immunity. Parasite Immunol. 2019 Mar;41(3):e12573. doi: 10.1111/pim.12573. Epub 2018 Aug 28. PMID 30019470
- [Result] Briggs J, Ategeka J, Kajubi R, Ochieng T, Kakuru A, Ssemanda C, Wasswa R, Jagannathan P, Greenhouse B, Rodriguez-Barraquer I, Kamya M, Dorsey G. Impact of Microscopic and Submicroscopic Parasitemia During Pregnancy on Placental Malaria in a High-Transmission Setting in Uganda. J Infect Dis. 2019 Jul 2;220(3):457-466. doi: 10.1093/infdis/jiz130. PMID 30891605
- [Result] Okiring J, Olwoch P, Kakuru A, Okou J, Ochokoru H, Ochieng TA, Kajubi R, Kamya MR, Dorsey G, Tusting LS. Household and maternal risk factors for malaria in pregnancy in a highly endemic area of Uganda: a prospective cohort study. Malar J. 2019 Apr 23;18(1):144. doi: 10.1186/s12936-019-2779-x. PMID 31014336
- [Result] Kakuru A, Jagannathan P, Kajubi R, Ochieng T, Ochokoru H, Nakalembe M, Clark TD, Ruel T, Staedke SG, Chandramohan D, Havlir DV, Kamya MR, Dorsey G. Impact of intermittent preventive treatment of malaria in pregnancy with dihydroartemisinin-piperaquine versus sulfadoxine-pyrimethamine on the incidence of malaria in infancy: a randomized controlled trial. BMC Med. 2020 Aug 10;18(1):207. doi: 10.1186/s12916-020-01675-x. PMID 32772921
- [Result] Savic RM, Jagannathan P, Kajubi R, Huang L, Zhang N, Were M, Kakuru A, Muhindo MK, Mwebaza N, Wallender E, Clark TD, Opira B, Kamya M, Havlir DV, Rosenthal PJ, Dorsey G, Aweeka FT. Intermittent Preventive Treatment for Malaria in Pregnancy: Optimization of Target Concentrations of Dihydroartemisinin-Piperaquine. Clin Infect Dis. 2018 Sep 14;67(7):1079-1088. doi: 10.1093/cid/ciy218. PMID 29547881
- [Result] Ategeka J, Kakuru A, Kajubi R, Wasswa R, Ochokoru H, Arinaitwe E, Yeka A, Jagannathan P, Kamya MR, Muehlenbachs A, Chico RM, Dorsey G. Relationships Between Measures of Malaria at Delivery and Adverse Birth Outcomes in a High-Transmission Area of Uganda. J Infect Dis. 2020 Aug 4;222(5):863-870. doi: 10.1093/infdis/jiaa156. PMID 32249917
- [Result] Roh ME, Kuile FOT, Rerolle F, Glymour MM, Shiboski S, Gosling R, Gutman J, Kakuru A, Desai M, Kajubi R, L'Ianziva A, Kamya MR, Dorsey G, Chico RM. Overall, anti-malarial, and non-malarial effect of intermittent preventive treatment during pregnancy with sulfadoxine-pyrimethamine on birthweight: a mediation analysis. Lancet Glob Health. 2020 Jul;8(7):e942-e953. doi: 10.1016/S2214-109X(20)30119-4. PMID 32562650
- [Derived] Vaaben AV, Levan J, Nguyen CBT, Callaway PC, Prahl M, Warrier L, Nankya F, Musinguzi K, Kakuru A, Muhindo MK, Dorsey G, Kamya MR, Feeney ME. In Utero Activation of Natural Killer Cells in Congenital Cytomegalovirus Infection. J Infect Dis. 2022 Sep 4;226(4):566-575. doi: 10.1093/infdis/jiac307. PMID 35876164
- [Derived] Hughes E, Wallender E, Kajubi R, Jagannathan P, Ochieng T, Kakuru A, Kamya MR, Clark TD, Rosenthal PJ, Dorsey G, Aweeka F, Savic RM. Piperaquine-Induced QTc Prolongation Decreases With Repeated Monthly Dihydroartemisinin-Piperaquine Dosing in Pregnant Ugandan Women. Clin Infect Dis. 2022 Aug 31;75(3):406-415. doi: 10.1093/cid/ciab965. PMID 34864925
- [Derived] Zehner N, Adrama H, Kakuru A, Andra T, Kajubi R, Conrad M, Nankya F, Clark TD, Kamya M, Rodriguez-Barraquer I, Dorsey G, Jagannathan P. Age-Related Changes in Malaria Clinical Phenotypes During Infancy Are Modified by Sickle Cell Trait. Clin Infect Dis. 2021 Nov 16;73(10):1887-1895. doi: 10.1093/cid/ciab245. PMID 33738485
- [Derived] Kakuru A, Roh ME, Kajubi R, Ochieng T, Ategeka J, Ochokoru H, Nakalembe M, Clark TD, Ruel T, Staedke SG, Chandramohan D, Havlir DV, Kamya MR, Dorsey G, Jagannathan P. Infant sex modifies associations between placental malaria and risk of malaria in infancy. Malar J. 2020 Dec 3;19(1):449. doi: 10.1186/s12936-020-03522-z. PMID 33272281

RESULTS

PARTICIPANT FLOW:
Groups:
- Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy: Women will be given SP (3 full strength tabs, 500 mg/25 mg) every four weeks times during pregnancy. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two drugs on day 1 (SP and placebo or DP and placebo) followed by one drug on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy
- Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy: Women will be given DP (3 full strength tabs, 40 mg/320 mg, given once a day for 3 consecutive days) every 4 weeks during pregnancy. In addition, placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two drugs on day 1 (SP and placebo or DP and placebo) followed by one drug on days 2 and 3 (DP or placebo). Two placebos will be used, one that mimics the appearance of SP and one that mimics the appearance of DP.
  Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Period: Overall Study
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Started | 391 | 391
Completed | 338 | 349
Not Completed | 53 | 42
Not completed — Lost to Follow-up | 31 | 19
Not completed — Withdrawal by Subject | 21 | 17
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy | Total
Number analyzed (Participants) | 391 | 391 | 782
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [19 to 27] | 23 [19 to 27] | 23 [19 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 391 | 391 | 782
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 391 | 391 | 782
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 391 | 391 | 782
Gestational age category (weeks) [Count of Participants; unit: Participants]
  12-16 weeks | 234 | 242 | 476
  >16-20 weeks | 157 | 149 | 306
Detection of malaria parasites by microscopy or qPCR [Count of Participants; unit: Participants] | 326 | 317 | 643

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Deliver With a Composite Adverse Birth Outcome
Description: Composite adverse birth outcome defined as any one of the following: 1) Low birth weight (< 2500 gm); 2) Preterm delivery (< 37 weeks gestational age); 3) Small for gestational age (< 10th percentile relative to an external growth reference)
Time Frame: Delivery
Population: Number of livebirths reported here. SP: 338 women followed through delivery resulting in 348 infants (10 twin sets). 9 mothers/infants excluded (4 spontaneous abortions, 5 stillbirths).
  DP: 349 women followed through delivery resulting in 352 infants (3 twin sets). 12 mothers and 13 infants excluded (10 spontaneous abortions, 3 stillbirths).
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 329 | 337
Participants | 60 | 54

2. Primary Outcome: Incidence of Malaria in Infants
Description: episodes per person year
Time Frame: Time at risk will begin at birth and end when study participants reaches 12 months of age or early study termination
Population: 339 live births included in the analyses for both groups.
Measure: Number; unit: episodes per person year
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 339 | 339
episodes per person year | 1.98 | 1.71

3. Primary Outcome: Mean Gestational Age in Weeks at Birth
Description: Gestational age in weeks determined by ultrasound dating (gold standard) and by the metabolic profiling outcome from biological specimens including placental tissue and placental blood.
Time Frame: At the time of delivery
Population: 339 live births included in the analyses for both groups.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 339 | 339
weeks | 39.4 (1.9) | 39.6 (1.6)

4. Secondary Outcome: Prevalence of Placental Malaria by Histology
Description: Any evidence of placental infection (parasites or pigment). Number of participants with placental tissue positive for malaria parasites or pigment.
Time Frame: Delivery
Population: analysis population is women who delivered and had histopathology results (i.e. some women who delivered did not have histopathology results)
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 322 | 331
Participants | 197 | 94

5. Secondary Outcome: Prevalence of Placental Parasitemia
Description: Proportion of placental blood samples positive for parasites by Loop-mediated isothermal amplification (LAMP) or microscopy
Time Frame: Delivery
Population: LAMP and microscopy performed for the number of participants reported in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 339 | 339
Participants
  LAMP: number analyzed (Participants) | 320 | 329
  LAMP | 71 | 7
  Microscopy: number analyzed (Participants) | 326 | 331
  Microscopy | 29 | 1

6. Secondary Outcome: Prevalence of Maternal Malaria
Description: Maternal blood positive for malaria parasites by microscopy.
Time Frame: Gestational age between 12-20 weeks (at study entry) up to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 336 | 342
Participants | 28 | 1

7. Secondary Outcome: Number of Participants With Adverse Events
Description: All grade 3 and 4 adverse events
Time Frame: Starting at the time of their first study drug administration, approximately gestational age between 12-20 weeks, up to one month post-delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 375 | 373
Participants | 54 | 43

8. Secondary Outcome: Prevalence of Anemia in Pregnant Women
Description: hemoglobin < 11 g/dL
Time Frame: as for outcome 7
Population: Number of women initiated on study drugs reported here.
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 375 | 373
Participants | 28 | 8

9. Secondary Outcome: Prevalence of Anemia in Infants
Description: Defined as the proportion with hemoglobin < 10 g/dL measure routinely at 12, 28, and 52 weeks of age. Number of cases per person year (PPY).
  This is a prevalence measure but are repeated measures during infancy. In other words we measured this outcome up to 3 times for each participant during infancy (at 12, 28 and 52 weeks of age).
Time Frame: Birth up to 12 months of age or early termination
Population: 339 live births included in the analyses for both groups.
Measure: Count of Units; unit: routine hemoglobin measurement
Units Other Than Participants: routine hemoglobin measurement
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 339 | 339
Number analyzed (routine hemoglobin measurement) | 878 | 892
routine hemoglobin measurement | 222 | 216

10. Secondary Outcome: Prevalence of Asymptomatic Parasitemia in Pregnant Women
Description: Proportion of routine monthly samples positive for parasites by microscopy and LAMP
Time Frame: as for outcome 7
Measure: Count of Units; unit: blood smears
Units Other Than Participants: blood smears
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 391 | 391
Number analyzed (blood smears) | 1687 | 1757
blood smears | 519 | 9

11. Secondary Outcome: Prevalence of Asymptomatic Parasitemia in Infants
Description: Proportion of routine monthly samples positive for parasites by microscopy and LAMP
Time Frame: Birth up to 12 months of age or early termination
Measure: Count of Units; unit: blood smears
Units Other Than Participants: blood smears
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 339 | 339
Number analyzed (blood smears) | 3879 | 3933
blood smears | 344 | 357

12. Secondary Outcome: Incidence of Complicated Malaria in Infants
Description: Complicated malaria defined as an episode of malaria with danger signs (any of the following: less than 3 convulsions over 24 h, inability to sit or stand, vomiting everything, unable to breastfeed or drink) or the meeting standardized criteria for severe malaria.
Time Frame: Birth up to 12 months of age or early termination
Population: 339 live births included in the analyses for both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 339 | 339
Participants | 44 | 24

13. Secondary Outcome: Incidence of Hospital Admissions in Infants
Description: Admission to the pediatric ward for any cause
Time Frame: Birth up to 12 months of age or early termination
Population: 339 live births included in the analyses for both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 339 | 339
Participants | 19 | 8

14. Secondary Outcome: Infant Mortality Rate
Description: Any deaths occurring after birth
Time Frame: Birth up to 12 months of age
Population: 339 live births included in the analyses for both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
Number analyzed (Participants) | 339 | 339
Participants | 9 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected following the initiation of study drugs through to 6 weeks postpartum.
Description: Adverse events were assessed and graded according to standardized criteria (National Institutes of Health, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0) at every visit to the study clinic.
  The number of participants at risk are all women that were enrolled, randomized, AND received at least 1 dose of study drugs.
Arm/Group | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy
All-Cause Mortality (participants affected / at risk) | 1/375 | 3/373
Serious Adverse Events (participants affected / at risk) | 11/375 | 19/373
Other Adverse Events (participants affected / at risk) | 341/375 | 341/373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy (N=375) | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy (N=373)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Congenital anomaly (Congenital, familial and genetic disorders) | 2 (2) | 10 (10) — Birthed infant with congenital anomaly
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Elevated Alanine Aminotransferase (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Altered mental status (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monthly Sulfadoxine-Pyrimethamine (SP) During Pregnancy (N=375) | Monthly Dihydroartemisinin-Piperaquine (DP) During Pregnancy (N=373)
Abdominal pain (General disorders) | 273 (822) | 282 (800)
Cough (General disorders) | 254 (603) | 268 (681)
Headache (General disorders) | 256 (586) | 237 (604)
Pyuria (Renal and urinary disorders) | 51 (63) | 59 (69)
Diarrhea (Gastrointestinal disorders) | 50 (62) | 49 (66)
Malaise (General disorders) | 48 (54) | 44 (52)
Vomitting (Gastrointestinal disorders) | 34 (44) | 35 (45)
Chills (General disorders) | 26 (27) | 24 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT02793622/Prot_SAP_000.pdf